CLINICAL TRIAL: NCT06009406
Title: Comparison of the Instantaneous Effects of Graston Technique and Static Stretching on Ankle Range of Motion and Vertical Jump Performance in Athletes
Brief Title: Comparison of the Effect of Graston Technique and Static Stretching in Athletes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Muğla Sıtkı Koçman University (Other)
Responsible Party: Principal Investigator, Fatih Ozden, Assistant Professor, Muğla Sıtkı Koçman University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: graston
Record Dates: First submitted 2023-08-19; First posted 2023-08-24 (Actual); Last update posted 2024-03-27 (Actual); Status verified 2024-03

CONDITIONS: Physical Therapy
MeSH Terms: interventions — Physical Therapy Modalities

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): This group will be applied to the soleus, gastrocnemius muscle and Achilles tendon with Graston, an instrumental myofascial mobilization technique, until they feel warmth in the skin and tonus relaxation in the target muscles. The persons treated with graston are applied at a 45° angle parallel to the muscle fibers for approximately 20 seconds. Immediately afterwards, the graston is applied to the muscles in a direction perpendicular to the same muscle fibers at a 45° angle for 20 seconds, resulting in a total treatment time of approximately 40 seconds. This results in an increase in temperature and tonus relaxation on the skin surface. In our study, the application will be performed for Gastarocnemius, Soleus muscle and Achilles tendon.
  Interventions: Other: Physiotherapy
- Control Group (Active Comparator): The control group will be subjected to 3 repetitions of passive stretching for 30 seconds for the same structures. The static stretching technique is a widely used method that lengthens muscle length by autogenic inhibition that stimulates the Golgi tendon organ. This technique involves passively stretching a specific antagonist muscle by placing it in a position of maximum stretch and holding it there for an extended period of time. Recommendations on the optimal length of time to hold this flexed position typically indicate that a 30-second hold, repeated 3 to 4 times, will provide the most beneficial results. 3 repetitions of passive stretching for 30 seconds will be applied to the same structures.
  Interventions: Other: Physiotherapy

INTERVENTIONS:
Other: Physiotherapy — This group will be applied to the soleus, gastrocnemius muscle and Achilles tendon with Graston, an instrumental myofascial mobilization technique, until they feel warmth in the skin and tonus relaxation in the target muscles. The control group will be subjected to 3 repetitions of passive stretching for 30 seconds for the same structures.

SUMMARY:
In our study, we aimed to compare the effects of both Graston technique and static stretching on ankle range of motion and vertical jump performance in the light of the literature. Our study will guide clinicians about the uncertainty in the application of Graston technique and static stretching to the gastrocnemius, soleus muscles and Achilles tendon and examine the applicability of Graston in athletes. It is also aimed to investigate the relationship between ankle range of motion and vertical jump performance.

ELIGIBILITY:
Inclusion Criteria:

* The participant has volunteered and agreed to participate with the consent form
* The participant is between the ages of 18-40
* The participant is able to perform the squat movement pattern
* Participant must be an active and licensed athlete

Exclusion Criteria:

* Health problem that will affect the participant's mobility or jump performance
* The participant has had a surgical procedure involving the ankle and knee in the last 6 months
* The presence of orthopedic injury of the participant's foot and ankle
* Participant has a neurological diagnosis
* The participant is pregnant
* The participant has an acute lower extremity injury

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-05-01 (Actual); Study Completion 2023-06-01 (Actual)

PRIMARY OUTCOMES:
Vertical Jump Test (VJT) | Change from Baseline VJT at 10 minutes
  It is a test with a high reliability rate for determining the athlete's jumping power. It was developed by Dr. Dudley Allen Sargent in 1921. In the test, a tape measure is attached to the wall. Stand upright with the feet shoulder-width apart and the dominant side facing the wall. Without lifting the feet off the floor, the highest point that can be reached on the tape measure is marked. Then, immediately after bending down by bending the hips and knees, the highest point that can be reached by jumping is asked to be marked by hand. The distance difference between both points is determined. The test is repeated three times and the best result is recorded in centimeters.
Universal Goniometric Measurement (UGM) | Change from Baseline UGM at 10 minutes
  The participant lies supine with the knee extended and the ankle hanging over the end of the table. Inversion, eversion, dorsi flexion and plantar flexion active ankle range of motion can be assessed using a goniometer. In the universal goniometric measurement, the 90-degree right angle between the 5th metatarsal and fibula is considered the starting position of the ankle at 0 degrees for dorsi and plantar flexion. Since the gastrocnemius covers two joints, the muscle should be relaxed by placing a thin pillow under the knees during the measurement. The pivot point of the goniometer is placed on the lateral malleolus. The fixed arm is held parallel to the lateral midline of the fibula. The movable arm follows the lateral midline of the 5th metatarsal bone. Care is taken to avoid inversion and eversion of the foot during measurement.

CONTACTS AND LOCATIONS:
Overall Officials: İsmail Uysal, PhD, Study Director — Muğla Sıtkı Koçman University
Locations (1):
- FizyoMove, Istanbul, Üsküdar, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No